CLINICAL TRIAL: NCT03442478
Title: The Performance of Digital Breast Tomosynthesis Compared to Conventional Mammography in Visualization and Characterization of Suspicious Breast Abnormalities
Brief Title: Comparison of Digital Breast Tomosynthesis to Conventional Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-0138-C
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2D/3D Tomosynthesis (Experimental): 2D/3D Tomosynthesis images will be obtained in addition to standard mammographic images.
  Interventions: Other: 2D/3D Tomosynthesis

INTERVENTIONS:
Other: 2D/3D Tomosynthesis

SUMMARY:
In March 2009, Health Canada approved Tomosynthesis for use in screening and diagnosis of breast cancer. The Tomosynthesis technology is designed as a complementary imaging model that is incorporated into the 2D Mammography system. This new imaging system has the capability to provide 2D, 3D and combination mode models. It consists of generating thin slice images that can be viewed individually as multiple images from the same breast. Tomosynthesis provides improved visibility of possible lesions within the breast. The study aims to compare the performance of Tomosynthesis to the conventional Digital Mammography in detecting and characterizing suspicious findings in subjects who will be having breast biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female of any race and ethnicity
* Following routine mammography imaging, subject is categorized as Breast Imaging Reporting and Data System (BI-RADS®) 4 or 5 because of calcifications / masses and architectural distortion will undergo study imaging within 30 days of routine imaging
* Subject will undergo 2D/3D digital breast tomosynthesis prior to biopsy

Exclusion Criteria:

* Subject unable or unwilling to undergo informed consent
* Subjects who are unable or unwilling to tolerate compression
* Subjects who are pregnant or who think they may be pregnant
* Subjects who are breast-feeding
* The subject is too large to be imaged on the large 24 x 30 cm detector

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Comparison of Tomosynthesis to Standard Digital Mammography | 2 years
  To compare the sensitivity, specificity, positive and negative predictive values of tomosynthesis to conventional digital mammography in visualization and characterization of suspicious abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Anabel Scaranelo, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, University Health Network, 610 University Ave., Toronto, Ontario, Canada